CLINICAL TRIAL: NCT01532323
Title: Oral Sphere: Salivary Markers and Food. A Prospective Study in Children Expressing Oral Disorders
Acronym: ORALISENS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2011.671
Record Dates: First submitted 2012-01-31; First posted 2012-02-14 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2013-09

CONDITIONS: Oral Disorder
Keywords: Oral disorders
MeSH Terms: conditions — Mouth Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral disorder children (Experimental): Oral disorder children aged 2 to 15 years
  Interventions: Other: Taking of saliva before and after gustatory stimulation
- Control group (Active Comparator): No oral disorder children aged 2 to 15 years
  Interventions: Other: Taking of saliva before and after gustatory stimulation

INTERVENTIONS:
Other: Taking of saliva before and after gustatory stimulation — Taking of saliva before and after gustatory stimulation (3 drops of citric acid 2.4 g / L)

SUMMARY:
In Human, the oral sphere is the first and main place where sensory stimuli are received and perceived. The phenomena occuring during food breakdown and sensory perception are complex and in this system saliva plays a major role.

In the neonatal period, severe digestive diseases require the cessation of all oral feeding and the use of enteral or parenteral nutrition for prolonged periods to ensure the growth and development of children while their disease is active. The early stages of sensory oral exposures and their consequences on the development of eating habits of these children are poorly documented. It is likely that the process of acquisition of preferences and eating habits is atypical because of a "bypass" of the oral sphere during the early stages of feeding. Thus, if not orally fed, children do not get exposed to a wide variety of tastes and textures in the first year of life, which may impact on their oral acceptance at a later age. These oral disorders (OD) are expressed by a refusal to eat, a heightened gag reflex, a refusal of certain consistencies and difficulties in chewing and swallowing. Few data are available on food typically accepted by these children.

Finally, oral sensory phenotypes of OD children (gustatory sensitivity ...) have not been described yet. It is likely that they may differ significantly from those of healthy (NOD).

In this context, a population of OD children is particularly interesting for studying the effects of the absence of these learning stages and their consequences in the development of sensory perception and eating habits.

The investigators formulate the hypothesis that the lack of exposure to a standard oral diet would modify the development of their "oro-sensory systems" including saliva.

Studying such a population is a great opportunity to assess the influence of non oral food exposures and diet on saliva characteristics.

Saliva has recently received attention as a potential easy to collect source of biomarkers in several conditions excluding OD.

The potential impact of OD on salivary composition has never been studied. Several studies linking saliva and perception or preferences have been conducted in the UMR CSGA (Unité Mixte de Recherche du Centre des Sciences du Goût et de l'Alimentation). They have already contributed to highlight the great inter-individual variability for a number of saliva markers and a change in saliva protein profiles in response to taste stimulation They also underlined the remarkable intra-stability for saliva flow and composition during a one year study.

This study intends to prove the concept that it is relevant to relate saliva characteristics to food intake behaviour or food habits The first hypothesis to be tested in this study is that salivary profiles (biological signatures) can discriminate two groups of children differing by their orality.

The second hypothesis to be tested is that these specific biological biological signatures may be correlated to certain food habits associated or not with oral disorders.

ELIGIBILITY:
Inclusion Criteria:

Oral disorder children group:

* Oral disorder children, of any etiology, defined as follows:

difficulty to wean the nutritional support within 50% of energy intake recommended by age oral more than 3 months of exclusive artificial feeding during the first 6 months of life

* Children aged 2 to 15 years
* Children with a maximum of 50% of their energy intake provided by the oral route (3 or 4 patients with 0% intake, defined as an internal control)
* Whose parents gave consent for study participation

No oral disorder children group:

* No oral disorder children
* whose parents signed an informed consent for the participation of their child to the study

Exclusion Criteria:

Oral disorder children group:

* Child refusing to participate
* Absence of parents consent
* Less than 3 months of artificial feeding during the first 6 months of life,
* Immunosuppressive medication that might interfere with the saliva composition,
* Children not covered by the social security

No oral disorder children group:

* Child refusing to participate
* Absence of parents consent
* History of or current enteral or parenteral feeding.
* Children not covered by the social security

No oral disorder children are matched to Oral disorder children on age and sex.

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2011-12; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Change in lipase, protease, amylase and lysosomal activity, metabolomic, proteomic or peptidic analysis on saliva samples at enrolment, and at months 3, 6, 9 and 12 | at enrolment, and at months 3, 6, 9 and 12

SECONDARY OUTCOMES:
change in enzyme activities, metabolomic, proteomic and peptidic analysis before and after acidic stimulation of saliva at enrolment, and at months 3, 6, 9 and 12. | at enrolment, and at months 3, 6, 9 and 12
Types of diet and eating habits questionnaire | at enrolment, 6 months and 12 months after enrolment
Evolution of lipase, protease, amylase and lysosomal activity and metabolomic, proteomic and peptidic analysis of saliva at enrolment, and at months 3, 6, 9 and 12. | at enrolment, and at months 3, 6, 9 and 12

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Gastroentérologie, hépatologie et nutrition Hopital Femme Mere Enfant, Bron, France

REFERENCES:
- [Result] Morzel M, Truntzer C, Neyraud E, Brignot H, Ducoroy P, Lucchi G, Canlet C, Gaillard S, Nicod F, Nicklaus S, Peretti N, Feron G. Associations between food consumption patterns and saliva composition: Specificities of eating difficulties children. Physiol Behav. 2017 May 1;173:116-123. doi: 10.1016/j.physbeh.2017.02.005. Epub 2017 Feb 6. PMID 28185876